CLINICAL TRIAL: NCT02241330
Title: Efficacy of Zn Biofortified Wheat in Improving Zn Status in Indian School Children With Low Zn Status: a Randomized Controlled Trial
Brief Title: Efficacy of Zn Biofortified Wheat in Improving Zn Status in Indian School Children With Low Zn Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: HarvestPlus (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Prof, Swiss Federal Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EK 2013-N-52
Record Dates: First submitted 2014-09-09; First posted 2014-09-16 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Zinc Deficiency
Keywords: Zinc; deficiency; biofortification; wheat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Placebo Comparator): Control wheat used for meal, level of zinc is usual
  Interventions: Dietary Supplement: Control
- fortification (Active Comparator): Fortification Wheat is fortified before testmeal administration. Zinc level is comparable to WHO recommendation
  Interventions: Dietary Supplement: Fortification
- Biofortified (Active Comparator): Biofortification Biofortified wheat is used for testmeal administration. Zinc concentration is around 30% higher than control
  Interventions: Dietary Supplement: Biofortified wheat

INTERVENTIONS:
Dietary Supplement: Biofortified wheat — Wheat was grown by foliar Zn application and is therefore biofortified
  Arms: Biofortified
Dietary Supplement: Fortification — Wheat flour is fortified before testmeal preparation
  Arms: fortification
Dietary Supplement: Control — wheat flour is used as control comparator.
  Arms: Control

SUMMARY:
The objective of this research is to test the efficacy of Zn biofortified wheat in increasing Zn status in Indian school children aged 6-12 y via a 6 month randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy

Exclusion Criteria:

* unhealthy

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 284 (Actual)
Dates: Start 2014-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change of plasma zinc values from baseline to endpoint and two months post intervention | day 0, random between day 0 and 6 month, 6 month and random between 6 months and 2 months post-intervention
  plasma zinc will be measured at baseline, midpoint (random sparse sampling), endpoint (6 months) and randomly within two months post-intervention

SECONDARY OUTCOMES:
Change in the Inflammation marker from baseline to the end of the intervention, as well as post-intervention | day 0, random during the intervention, month 6, and random 2 months post intervention
  CRP will be measured at baseline, midpoint (random sparse sampling), endpoint (end of intervention) and randomly within two months post-intervention
Change in the chronic inflammation marker from baseline to 6 months and 2 month post intervention | day 0, random during the intervention, month 6, and random 2 months post intervention
  AGP will be measured at baseline, midpoint (random sparse sampling), endpoint (6 months)and randomly within two months post-intervention
Change in Iron status from baseline to the end of the intervention and 2 months post-intervention | day 0, random during the intervention, month 6, and random 2 months post intervention
  Hb will be measured at baseline, midpoint (random sparse sampling), endpoint (6 months) and randomly within two months post-intervention
Change in Iron status from baseline to the end of intervention, and within two months post-intervention | day 0, random during the intervention, month 6, and random 2 months post intervention
  Serum ferritin will be measured at baseline, midpoint (random sparse sampling), endpoint and randomly within two months post-intervention
New Zn biomarkers | day 0, random during the intervention, month 6, and random 2 months post intervention
  new potential zn biomarkers will be measured in whole blood and plasma at baseline, midpoint (random sparse sampling), endpoint and randomly within two months post-intervention
New potential Zn biomarkers in buccal cells | day 0, random during the intervention, month 6, and random 2 months post intervention
  MT RNA transcript in buccal cells will be measured at baseline, midpoint (random sparse sampling), endpoint
Characterization of gut microflora | baseline, endpoint (6 months)
  Characterization of microflora will be done in a subsamples of children (taken randomly), at baseline and at the end of feeding (6 months)
Anthropometry | baseline (day 0), endpoint (6 months)
  anthropometry, such as height, weight will be measured at baseline and endpoint of the study
morbidity | throughout the study
  morbidity, mainly diarrhea and pneumonia episodes, will be recorded throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Zimmermann, Prof Dr med, Principal Investigator — ETHZ; Anura V Kurpad, Prof MD PhD, Principal Investigator — St John's Research Institute, Bangalore
Locations (1):
- St John's Research Institute, Bangalore, Karnataka, India

REFERENCES:
- [Derived] Signorell C, Kurpad AV, Pauline M, Shenvi S, Mukhopadhyay A, King JC, Zimmermann MB, Moretti D. The Effect of Zinc Biofortified Wheat Produced via Foliar Application on Zinc Status: A Randomized, Controlled Trial in Indian Children. J Nutr. 2023 Oct;153(10):3092-3100. doi: 10.1016/j.tjnut.2023.08.013. Epub 2023 Aug 25. PMID 37633331
- See also: HarvestPlus website — http://www.harvestplus.org
- See also: St John's Research Institute website — http://www.sjri.res.in/